CLINICAL TRIAL: NCT03660241
Title: A PHASE 1, NON-RANDOMIZED, OPEN-LABEL, SINGLE-DOSE STUDY TO EVALUATE THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF PF-04965842 IN SUBJECTS WITH RENAL IMPAIRMENT AND IN HEALTHY SUBJECTS WITH NORMAL RENAL FUNCTION
Brief Title: A Renal Impairment Study for PF-04965842
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B7451021; 2018-002865-20 (EudraCT Number)
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — abrocitinib

STUDY DESIGN:
Intervention Model Description: Part 1 will be conducted. The 8 subjects from the renal impaired group will be recruited before recruiting the 8 subjects without renal impairment function in Part 1. After statistical evaluation of results from Part 1, Part 2 may be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-04965842 (Experimental): PF 04965842 is an oral selevtive janus kinase (JAK) 1 inhibitor
  Interventions: Drug: PF-04965842

INTERVENTIONS:
Drug: PF-04965842 — PF 04965842 is a janus kinase (JAK) 1 inhibitor that is currently being developed for the treatment of atopic dermatitis (AD).

SUMMARY:
This study is a phase 1 non-randomized, open-label, single-dose, parallel-group study of PF 04965842 in subjects with severe renal impairment and subjects without renal impairment (Part 1) and in subjects with moderate renal impairment (Part 2).

DETAILED DESCRIPTION:
This is a Phase 1 non randomized, open label, single dose, parallel cohort, multisite study to investigate the effect of renal impairment on the pharmacokinetics, safety and tolerability of PF-04965842 after a single 200 mg oral dose. Subjects will be selected and categorized into normal renal function or renal impairment groups based on their estimated glomerular filtration rate. Part 1: A total of approximately16 subjects will be enrolled; approximately 8 subjects with severe renal impairment and approximately 8 with normal renal function. After statistical evaluation of results from Part 1, Part 2 may be conducted and approximately 8 subjects with moderate renal impairment will be enrolled. The total duration of participation from the Screening Visit to Day 4 will be a maximum of 31 days and from the Screening Visit to Follow-up Contact/Visit will be a maximum of 67 days.

ELIGIBILITY:
Inclusion Criteria:

* Breath alcohol test at Screening and Day -1 must be negative.
* Body mass index (BMI) of ≥ 17.5 to ≤ 40.0 kg/m2; and a total body weight >50 kg (110 lb).

Additional inclusion criteria for subjects with renal impairment:

* Meet the following eGFR criteria during the screening period based on the MDRD equation:

  * Severe renal impairment: eGFR <30 mL/min, but not requiring hemodialysis.
  * Moderate renal impairment (Part 2 only): eGFR ≥30 mL/min and <60 mL/min.
* Any form of renal impairment except acute nephritic syndrome (subjects with history of previous nephritic syndrome but in remission can be included).
* Stable concomitant drug regimen.

Exclusion Criteria:

* Renal transplant recipients.
* Urinary incontinence without catheterization.
* Subjects with clinically significant infections within the past 3 months (for example, those requiring hospitalization, or as judged by the Investigator), evidence of any infection (including influenza) within the past 7 days prior to baseline, history of disseminated herpes simplex infection or recurrent or disseminated herpes zoster.
* Subjects with a malignancy or with a history of malignancy, with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* History of or current positive results for human immunodeficiency virus, Hepatitis B, Hepatitis C.

Additional exclusion criteria for subjects with renal impairment:

* Subjects requiring hemodialysis and peritoneal dialysis.
* Screening BP ≥ 180 mm Hg (systolic) or ≥ 110 mm Hg (diastolic).
* Screening supine 12-lead ECG demonstrating QTcF >470 msec or a QRS interval >120 msec.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (3):
  - University of Miami Division of Clinical Pharmacology, Miami, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
- Brussels Clinical Research Unit, Brussels, Be-bru, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wang EQ, Le V, Winton JA, Tripathy S, Raje S, Wang L, Dowty ME, Malhotra BK. Effects of Renal Impairment on the Pharmacokinetics of Abrocitinib and Its Metabolites. J Clin Pharmacol. 2022 Apr;62(4):505-519. doi: 10.1002/jcph.1980. Epub 2022 Feb 15. PMID 34637151
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451021

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Renal Function: Participants were selected and categorized into the normal renal function group with the estimated glomerular filtration rate (eGRF) based on Modification of Diet in Renal Disease (MDRD) formula >=90 mL/min on Day -1. Participants received a single 200 mg oral dose of PF-04965842 on Day 1 after a fast of at least 10 hours.
- Moderate Renal Impairment: Participants were selected and categorized into the moderate renal impairment group with the estimated glomerular filtration rate (eGRF) based on Modification of Diet in Renal Disease (MDRD) formula >=30 and <60 mL/min on Day -1. Participants received a single 200 mg oral dose of PF-04965842 on Day 1 after a fast of at least 10 hours.
- Severe Renal Impairment: Participants were selected and categorized into the severe renal impairment group with the estimated glomerular filtration rate (eGFR) based on Modification of Diet in Renal Disease (MDRD) formula <30 mL/min on Day -1 and not requiring dialysis. Participants received a single 200 mg oral dose of PF-04965842 on Day 1 after a fast of at least 10 hours.
Period: Overall Study
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Started | 8 | 7 | 8
Completed | 8 | 7 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment | Total
Number analyzed (Participants) | 8 | 7 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (4.71) | 65.7 (8.34) | 61.0 (14.46) | 62.0 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 7
  Male | 6 | 3 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 4 | 12
  Not Hispanic or Latino | 4 | 3 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 6 | 6 | 7 | 19
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for PF-04965842
Description: Maximum observed plasma PF-04965842 concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8
nanogram per milliliter (ng/mL) | 1174 (56) | 1626 (31) | 1164 (80)
Statistical Analysis 1: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test: the moderate renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 138.49, 90% CI 2-sided [93.74 to 204.61]
Statistical Analysis 2: Comparison: Normal Renal Function vs Severe Renal Impairment; Test: the severe renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 99.11, 90% CI 2-sided [57.30 to 171.43]

2. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) for PF-04965842
Description: Area under the plasma PF-04965842 concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose.
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7
nanogram*hour per milliliter (ng*hr/mL) | 4827 (65) | 8828 (37) | 5855 (73)
Statistical Analysis 1: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test: the moderate renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 182.91, 90% CI 2-sided [117.09 to 285.71]
Statistical Analysis 2: Comparison: Normal Renal Function vs Severe Renal Impairment; Test: the severe renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 121.32, 90% CI 2-sided [68.32 to 215.41]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for PF-06471658 (M1)
Description: Maximum observed plasma concentration for active metabolite, PF-06471658 (M1).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose.
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8
nanogram per milliliter (ng/mL) | 193.7 (54) | 192.8 (65) | 325.0 (81)
Statistical Analysis 1: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test: the moderate renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 99.51, 90% CI 2-sided [59.80 to 165.57]
Statistical Analysis 2: Comparison: Normal Renal Function vs Severe Renal Impairment; Test: the severe renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 167.79, 90% CI 2-sided [97.20 to 289.64]

4. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) for PF-06471658 (M1)
Description: Area under the plasma concentration-time profile from time 0 extrapolated to infinite time for active metabolite, PF-06471658 (M1).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose.
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8
nanogram*hour/milliliter (ng*hr/mL) | 872.6 (44) | 1346 (43) | 2505 (45)
Statistical Analysis 1: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test: the moderate renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 154.22, 90% CI 2-sided [105.11 to 226.26]
Statistical Analysis 2: Comparison: Normal Renal Function vs Severe Renal Impairment; Test: the severe renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 287.06, 90% CI 2-sided [196.72 to 418.89]

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for PF-07055087 (M2)
Description: Maximum observed plasma concentration for active metabolite, PF-07055087 (M2).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose.
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8
nanogram per milliliter (ng/mL) | 241.3 (34) | 331.6 (21) | 429.3 (28)
Statistical Analysis 1: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test: the moderate renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 137.43, 90% CI 2-sided [106.82 to 176.81]
Statistical Analysis 2: Comparison: Normal Renal Function vs Severe Renal Impairment; Test: the severe renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 177.92, 90% CI 2-sided [135.91 to 232.92]

6. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) for PF-07055087 (M2)
Description: Area under the plasma concentration-time profile from time 0 extrapolated to infinite time for active metabolite, PF-07055087 (M2).
Time Frame: 0 (pre-dose), and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose.
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8
nanogram*hour per milliliter (ng*hr/mL) | 1476 (31) | 3981 (38) | 8433 (25)
Statistical Analysis 1: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test: the moderate renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 269.78, 90% CI 2-sided [196.61 to 370.18]
Statistical Analysis 2: Comparison: Normal Renal Function vs Severe Renal Impairment; Test: the severe renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 571.43, 90% CI 2-sided [447.27 to 730.05]

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Adverse events (AEs): any untoward medical occurrence in a clinical investigation subject administered a product or medical device, without regard to causality. Treatment-emergent AEs (TEAEs): AEs which occurred for the first time during the effective duration of treatment or AEs that increased in severity during treatment. Serious AEs (SAEs) were any untoward medical occurrence at any dose that resulted in death; was life-threatening; required inpatient hospitalization or caused prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions). AEs included SAEs and non-serious AEs. Treatment-related TEAEs were any untoward medical occurrence attributed to study treatment. Causality to study treatment was determined by the investigator.
Time Frame: Baseline up to Follow-Up (Day 36)
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8
Participants
  All-causality | 1 | 1 | 0
  Treatment-related | 0 | 1 | 0

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Protocol-required safety laboratory assessments included chemistry, hematology, and urinalysis (and microscopy, if needed). Each parameter was evaluated against commonly used and widely accepted criteria.
Time Frame: Baseline, post-dose on Day 1, Day 2 and Day 4.
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8
Participants | 6 | 6 | 8

9. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Values
Description: Vital sign data included blood pressure and pulse rate. Clinical significance was assessed by the investigator.
Time Frame: Day 1 (pre-dose) and Day 4
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8
Participants | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Values
Description: Clinical significance of ECG data was assessed by the investigator.
Time Frame: Baseline, post-dose on Day 1 and on Day 4
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8
Participants | 0 | 0 | 0

11. Post Hoc Outcome: Unbound Maximum Observed Plasma Concentration (Cmax,u) of the Active Moiety
Description: The unbound maximum observed plasma concentration for active moiety, calculated as the sum of unbound Cmax for PF-04965842 and active metabolites, PF-06471658 (M1) and PF-07055087 (M2), adjusted for the relative potencies of the metabolites.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose.
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar (nM)
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8
nanomolar (nM) | 2099 (38) | 2810 (20) | 2718 (41)
Statistical Analysis 1: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test: the moderate renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 133.87, 90% CI 2-sided [102.45 to 174.92]
Statistical Analysis 2: Comparison: Normal Renal Function vs Severe Renal Impairment; Test: the severe renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 129.49, 90% CI 2-sided [92.86 to 180.57]

12. Post Hoc Outcome: Unbound Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf,u) of the Active Moiety
Description: The unbound area under the plasma concentration-time profile from time 0 extrapolated to infinite time for active moiety, calculated as the sum of unbound AUCinf for PF-04965842 and active metabolites, PF-06471658 (M1) and PF-07055087 (M2), adjusted for the relative potencies of the metabolites.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose.
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar*hour (nM*hr)
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7
nanomolar*hour (nM*hr) | 9955 (40) | 20920 (28) | 28940 (23)
Statistical Analysis 1: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test: the moderate renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 210.20, 90% CI 2-sided [154.60 to 285.80]
Statistical Analysis 2: Comparison: Normal Renal Function vs Severe Renal Impairment; Test: the severe renal impairment group; Reference: the normal renal function group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of adjusted geometric means = 290.68, 90% CI 2-sided [217.39 to 388.69]

ADVERSE EVENTS:
Time Frame: Baseline up to Follow-Up (Day 36)
Arm/Group | Normal Renal Function | Moderate Renal Impairment | Severe Renal Impairment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 1/7 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function (N=8) | Moderate Renal Impairment (N=7) | Severe Renal Impairment (N=8)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT03660241/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT03660241/SAP_001.pdf